CLINICAL TRIAL: NCT03066583
Title: Prospective, Randomised, Double Blinded Trial Comparing Effectiveness of Platelet Rich Plasma or Placebo in a Primary Meniscal Tear Treatment
Brief Title: Effectiveness of Trephination With Platelet Rich Plasma or Placebo in a Primary Meniscal Tear Treatment
Acronym: Prolotherapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Rafał Kamiński, Deputy Chair of Division, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 501-1-07-18-15
Record Dates: First submitted 2016-10-21; First posted 2017-02-28 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Meniscus Lesion
Keywords: meniscus repair; platelet rich plasma
MeSH Terms: interventions — Trephining

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trephination with placebo (Placebo Comparator): meniscal repair with trephination and placebo
  Interventions: Biological: trephination with placebo
- trephination with platelet rich plasma (Experimental): meniscal repair with trephination and platelet rich plasma
  Interventions: Biological: trephination with platelet rich plasma

INTERVENTIONS:
Biological: trephination with placebo — trephination under US guidance and placebo injection
  Arms: trephination with placebo
Biological: trephination with platelet rich plasma — trephination under US guidance and platelet rich plasma injection
  Arms: trephination with platelet rich plasma

SUMMARY:
This study will compare meniscal healing augmented or without augmentation with platelet rich plasma in primary meniscal tear treatment (prolotherapy). The assessments will include validated, disease specific, patient oriented outcome measures. Results of this study will help ascertain whether platelet rich plasma may improve meniscal healing rates.

DETAILED DESCRIPTION:
The role of meniscal in the knee integrity is pivotal and lack or partial role of the meniscus increases rate of joint degeneration. Partial meniscal removal is the most popular procedure and meniscal repair remain in minority of arthroscopic surgeries. As criteria of inclusion to meniscal repair are very rough, still success rates of meniscal repair remain in the 60-80% range for isolated repairs. This rate is greater when performed with ACL reconstruction. The investigators believe that augmentation with platelet rich plasma as prolotherapy ill induce healing without the need for arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Complete horizontal 10 mm in length
* Tear located in the vascular/avascular portion of the meniscus (chronic horizontal tear on MR)
* Single tear of the medial and/or lateral meniscus
* Skeletally mature patients 18-70 years of age

Exclusion Criteria:

* discoid meniscus
* arthritic changes (Kellgren Lawrence scale >2) or axial leg deformity (valgus > 6 deg)
* inflammatory diseases (i.e. rheumatoid arthritis)
* concominant chondral defects (> 2 ICRS)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-01; Primary Completion 2019-01 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Assessment of meniscal healing by MR scanning | by 1 year
  The primary outcome measures will be assessment of meniscal healing integrity by MR scanning

SECONDARY OUTCOMES:
Visual Analog Scale | 12 weeks, 6months, 1year post procedure
  Pain Visual Analog Scale.
Knee injury and Osteoarthritis Outcome Score scale | 12 weeks, 6months, 1year post procedure
  Knee injury and Osteoarthritis Outcome Score
International Knee Documentation Committee - Subjective Knee Evaluation Form | 12 weeks, 6months, 1year post procedure
  International Knee Documentation Committee - Subjective Knee Evaluation Form

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Kaminski, Principal Investigator — PCME, Otwock, Poland
Locations (1):
- Department of Orthopaedics and Traumatology, Postgraduate Center for Medical Education, Professor A. Gruca Teaching Hospital, Otwock, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided